CLINICAL TRIAL: NCT06638931
Title: Phase II Basket Study to Evaluate the Tissue-agnostic Efficacy of Anti-Programmed Cell Death Protein 1 (Anti-PD1) Monoclonal Antibody in Patients With Advanced Rare Tumors
Brief Title: Agnostic Therapy in Rare Solid Tumors
Acronym: ANTARES
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Principal Investigator, Paulo Marcelo Gehn Hoff, Full Professor of Clinical Oncology in the Department of Radiology and Oncology at FMUSP (University of São Paulo Medical School)., Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP4021/2023; 68590423.0.1001.0068 (Registry Identifier: Certificate of Ethical Review Submission); 01.23.0265.00 (Other Grant/Funding Number: FINEP)
Record Dates: First submitted 2024-10-03; First posted 2024-10-15 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Urachal Cancer; Parathyroid Carcinoma; Fibrolamellar Carcinoma; Angiosarcoma; Secretory Carcinoma of Breast; Anal Neoplasms; Metaplastic Breast Carcinoma; Translocation Renal Cell Carcinoma; Carcinosarcoma; Small Intestine Neoplasms; Cholangiocarcinoma; Sertoli-Leydig Cell Tumor; Adenoid Cystic Carcinoma; Mesothelioma; Neuroblastoma; Adrenal Gland Neoplasms; Penile Neoplasms; Apocrine Carcinoma; Fibrosarcoma; Cancer of Unknown Primary; Hemangioblastoma; Thyroid Neoplasms; Hepatoblastoma; Fallopian Tube Neoplasms; Leiomyosarcoma; Vaginal Neoplasms; Neurofibrosarcoma; Gallbladder Neoplasms; Osteosarcoma; Biliary Tract Neoplasms; Clear Cell Endometrial Cancer; Yolk Sac Tumor; Vulvar Neoplasms; Kaposi Sarcoma; Ovarian Epithelial Cancer; Soft Tissue Sarcoma; Urethral Neoplasms; Granulosa Cell Tumor; Primitive Neuroectodermal Tumor; Neuroendocrine Tumors; Trophoblastic Tumor
Keywords: Urachal Adenocarcinoma; Parathyroid Carcinoma; Nasopharyngeal Epithelial Tumors; Fibrolamellar Carcinoma; Angiosarcoma; Secretory Breast Carcinoma; Anal Cancer; Metaplastic Breast Carcinoma; Chromophobe Renal Carcinoma; Carcinosarcoma; Small Intestine Cancer; Cholangiocarcinoma; Sertoli-Leydig Cell Tumors; Non-Squamous Cervical Neoplasm; Tracheal Epithelial Tumors; Non-Adenoid Cystic Salivary Tumors; Mesothelioma; Neuroblastoma; Adrenal Neoplasm; Penile Cancer; Apocrine Carcinoma; Fibrosarcoma; Cancer of Unknown Primary; Hemangioblastoma; Thyroid Cancer; Hepatoblastoma; Fallopian Tube Cancer; Leiomyosarcoma; Vaginal Cancer; Neurofibrosarcoma; Gallbladder Cancer; Osteosarcoma; Biliary Tract Cancer; Clear Cell Endometrial Cancer; Yolk Sac Tumor; Non-Squamous Bladder Cancer; Vulvar Cancer; Kaposi Sarcoma; Ovarian Epithelial Cancer; Soft Tissue Sarcoma; Urethral Cancer; Granulosa Cell Tumor; Adenoid Cystic Carcinoma; Primitive Neuroectodermal Tumor; Neuroendocrine Tumors; Trophoblastic Tumor
MeSH Terms: conditions — Urachal cancer; Parathyroid Neoplasms; Fibrolamellar hepatocellular carcinoma; Hemangiosarcoma; Secretory breast carcinoma; Anus Neoplasms; Carcinosarcoma; Cholangiocarcinoma; Sertoli-Leydig Cell Tumor; Carcinoma, Adenoid Cystic; Mesothelioma; Neuroblastoma; Adrenal Gland Neoplasms; Penile Neoplasms; Fibrosarcoma; Hemangioblastoma; Thyroid Neoplasms; Hepatoblastoma; Fallopian Tube Neoplasms; Leiomyosarcoma; Vaginal Neoplasms; Neurofibrosarcoma; Gallbladder Neoplasms; Osteosarcoma; Biliary Tract Neoplasms; Endodermal Sinus Tumor; Vulvar Neoplasms; Sarcoma, Kaposi; Carcinoma, Ovarian Epithelial; Sarcoma; Urethral Neoplasms; Granulosa Cell Tumor; Neuroectodermal Tumors, Primitive; Neuroendocrine Tumors; Trophoblastic Neoplasms; Urachal adenocarcinoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: The study aims to evaluate the efficacy of the anti-PD1 monoclonal antibody, nivolumab, in the treatment of patients with advanced or metastatic rare malignant neoplasms. This study will be conducted as a single-arm trial, including patients who have a Combined Positive Score (CPS) of 10 or greater and who have demonstrated progression on standard treatment. Participants will be monitored to determine their response to treatment and any adverse effects associated with the use of nivolumab. The expectation is to provide evidence regarding the efficacy of this immunotherapeutic agent in a difficult-to-treat population, contributing to the advancement of therapeutic options available for these patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single-Arm Efficacy Study (Experimental): Treatment will be administered with intravenous nivolumab at a dose of 480 mg every 4 weeks. Treatment will continue until limiting toxicity, disease progression, or for a maximum of 12 months as maintenance if the individual achieves stable disease, partial response, or complete response.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — The intervention consists of administering Nivolumab 480 mg intravenously every 4 weeks, with a +5 day window for postponement but not for advancement of treatment. Treatment will continue until limiting toxicity, disease progression, or for a maximum period of 12 months (13 cycles) as maintenance therapy, provided the patient maintains stable disease, a partial response, or a complete response. Patients who are off treatment for more than 56 days (2 cycles) due to Nivolumab-related toxicities or other clinical issues will be discontinued from the protocol.
  After 12 months of treatment or in the event of study discontinuation for any reason, patients will be followed by the research team via telephone every 60 days, with a +/- 7 day window, until death.

SUMMARY:
The ANTARES study is a phase II basket trial designed to evaluate the tissue-agnostic efficacy of the monoclonal anti-PD1 antibody, nivolumab, in patients with advanced or metastatic rare tumors.

The study aims to treat rare malignancies with PD-L1 expression (CPS ≥ 10), regardless of the tumor's tissue type or location. Patients who have not responded to standard treatments will be included, and treatment will last for up to 12 months. The study will assess objective response, progression-free survival, and biomarkers such as PD-L1, ctDNA, and microvesicles, in a multicenter collaborative effort to provide innovative therapeutic options for this underrepresented population

DETAILED DESCRIPTION:
The ANTARES study is a phase II "basket" trial designed to evaluate the tissue-agnostic efficacy of the monoclonal anti-PD1 antibody, nivolumab, in patients with advanced or metastatic rare tumors. A "basket" trial is an innovative type of clinical trial where patients with different types of cancers, but sharing a common molecular feature (in this case, PD-L1 expression), are treated with the same therapy, regardless of the tumor's site of origin. This approach allows for the evaluation of treatments targeting specific molecular characteristics, independent of the primary cancer type.

Rare tumors, as defined by the World Health Organization (WHO), have an incidence of fewer than six cases per 100,000 people per year. Although each rare cancer type is individually uncommon, collectively they account for 25-30% of all malignancies and are often underrepresented in clinical trials due to recruitment challenges and limited funding. As a result, patients with rare cancers generally have a poorer prognosis compared to those with more common tumors.

In this study, patients with advanced or refractory rare malignancies expressing PD-L1, with a combined positive score (CPS) of ≥10, will be treated with nivolumab. Treatment will be administered until disease progression or for a maximum duration of 12 months, aiming to assess the efficacy and safety of this tissue-agnostic immunotherapy approach. Efficacy will be measured according to RECIST v1.1 criteria, with objective response as the primary endpoint. Additionally, the study will assess response biomarkers, including PD-L1, circulating tumor DNA (ctDNA), and microvesicles, to better understand the correlation between biomarker expression and clinical outcomes.

This multicenter trial, with an estimated duration of four years, will be conducted at Institute of Cancer of the State of São Paulo (ICESP) and other partner institutions. The study aims to overcome existing barriers in rare cancer treatment by offering an innovative approach that explores the potential of personalized therapies based on molecular characteristics, rather than the tumor's primary site

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older.
2. Patients with immunohistochemistry for PD-L1 with a combined positive score (CPS) of 10 or higher.
3. Patients with progression or intolerance to already approved and accessible treatments for the specific neoplasm and population.
4. Documented disease progression radiologically after the last routine treatment.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Measurable lesion per RECIST v1.1. Lesions previously treated with radiotherapy can only be used as target lesions if they are confirmed to be progressing by imaging before enrollment.
7. Male participants must meet at least one of the following conditions:

   1. Considered infertile;
   2. No fertile partner;
   3. Has a fertile partner who agrees to follow contraceptive guidance throughout the study period and for at least 6 months after the last dose of Nivolumab;

      and
   4. Agrees to abstain from sperm donation throughout the study period and for at least 6 months after the last dose of Nivolumab.
8. Female participants must meet at least one of the following conditions:

   1. Considered infertile;
   2. Agrees to follow contraceptive guidance throughout the study period and for at least 6 months after the last dose of Nivolumab;
9. Estimated life expectancy greater than 12 weeks, as determined by the investigator or delegated sub-investigator.
10. Preserved organ functions defined by:

    * Absolute neutrophil count ≥ 1,000;
    * Hemoglobin ≥ 8.0 g/dL (patients may receive transfusions to reach this level);
    * Platelet count ≥ 100,000;
    * Total bilirubin ≤ 1.5 × Upper Limit of Normal (ULN), or ≤ 3.0 × ULN for patients with Gilbert's syndrome;
    * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN in the presence of liver metastases);
    * Creatinine clearance > 30 mL/min (estimated by Cockcroft-Gault).
11. Diagnosis of rare cancer (List I) confirmed by histopathological examination, with the possibility of including other types of rare tumors (incidence of less than 6 in every 100,000) after careful evaluation and approval by the study board.

    * List I:

      * Urachal adenocarcinoma
      * Parathyroid carcinoma
      * Nasopharyngeal epithelial tumors
      * Fibrolamellar carcinoma of any primary site
      * Angiosarcoma of any primary site
      * Secretory breast carcinoma
      * Anal cancer
      * Metaplastic breast carcinoma
      * Chromophobe renal carcinoma, Microphthalmia-associated Transcription Factor (MiT) family translocation renal carcinoma; renal carcinoma with Fumarate Hydratase (FH) or Succinate Dehydrogenase (SDH) deficiency
      * Carcinosarcoma of any primary site
      * Small intestine cancer
      * Cholangiocarcinoma
      * Sertoli-Leydig cell tumors
      * Cervical cancer of non-epidermoid histology
      * Tracheal epithelial tumors
      * Non-cystadenoma salivary gland tumors
      * Mesothelioma of any site
      * Neuroblastoma
      * Adrenal cancer
      * Penile cancer
      * Apocrine carcinoma
      * Fibrosarcoma of any primary site
      * Cancer of unknown primary site
      * Hemangioblastoma of any primary site
      * Thyroid cancer
      * Hepatoblastoma
      * Fallopian tube cancer
      * Leiomyosarcoma of any primary site
      * Vaginal cancer
      * Neurofibrosarcoma of any primary site
      * Gallbladder cancer
      * Osteosarcoma of any primary site
      * Bile duct cancer
      * Clear cell endometrial carcinoma
      * Yolk sac tumor of any primary site
      * Non-epidermoid bladder cancer
      * Vulvar cancer
      * Kaposi's sarcoma
      * Epithelial ovarian cancer
      * Soft tissue sarcoma
      * Urethral cancer
      * Granulosa cell tumor of any primary site
      * Cystadenoma carcinoma
      * Primitive neuroectodermal tumor of any primary site
      * Pure or mixed neuroendocrine tumors with neuroendocrine component
      * Trophoblastic tumor

Exclusion Criteria

1. Previous treatment lines with immunotherapy (immune checkpoint inhibitors).
2. Pregnant or breastfeeding individuals.
3. Limiting comorbidity, in the opinion of the investigator.
4. Active infection.
5. Major surgery within the last 4 weeks.
6. Functional class II or greater heart failure.
7. Myocardial infarction or stroke within the last 6 months.
8. History of pulmonary fibrosis or pneumonitis.
9. Autoimmune diseases, except for patients with vitiligo and/or controlled thyroid/hypothyroidism without the use of immunosuppressors.
10. Second invasive primary tumor diagnosed in the last 3 years and/or with active disease, except for localized skin tumors (non-melanoma) that have been treated with curative intent.
11. Patients with prolonged QT interval.
12. Uncontrolled Central Nervous System (CNS) metastases. Patients who have previously received local treatment, such as radiotherapy, will be eligible if clinical and radiological stability is demonstrated in the 2 weeks prior to the start of treatment. Patients must not be using corticosteroids for managing CNS disease.
13. Presence of meningeal carcinomatosis.
14. Worsening renal and liver function in the 14 days prior to enrollment.
15. History of solid organ transplantation with or without immunosuppression.
16. Patients with untreated acquired immunodeficiency. Immunocompromised patients may be included as long as they do not have active opportunistic disease and/or active infection, after thorough clinical evaluation by the investigator or sub-investigator. HIV-positive patients must have documented undetectable viral load prior to inclusion.
17. Chronic use of corticosteroids at doses greater than 10 mg/day of prednisone or equivalent. Patients with adrenal insufficiency of non-autoimmune etiology (e.g., previous bilateral adrenalectomy) may be included if they are clinically compensated with 10 mg/day of prednisone or equivalent or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 2 years
  Overall survival (in months) of patients with advanced or metastatic rare malignancies and CPS ≥ 10 following disease progression after prior treatments while receiving the anti-PD1 antibody Nivolumab.
Primary Endpoint | 2 years
  The primary outcome of the study is the disease control rate (DCR) based on imaging, considering the best response to treatment. A response rate of 5% will be considered non-promising, and a response rate of 25% will be considered promising. The study follows Simon's two-stage design, with type I error (alpha) set at 0.05 and type II error (beta) at 0.10. In the first stage, if at least 1 out of the first 9 participants achieves disease control (stable disease, partial response, or complete response), 16 additional participants will be recruited for the second stage.
  The study will be deemed positive if at least 3 out of 25 participants achieve disease control (partial response, complete response, or stable disease). A 10% drop-out rate (3 participants) is anticipated, bringing the maximum total recruitment to 28 participants.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 2 years
  Percentage of patients with a tumor size reduction, measured according to RECIST criteria.
Subgroup Analysis Based on PD-L1 Expression and CPS: | 2 years
  PD-L1 Expression: Proportion of patients showing PD-L1 positivity. CPS Subgroups: Proportion of patients with CPS between 10-20 and those with CPS > 20.
Correlation of Clinical Outcomes with Biomarker Assessments | 2 years
  Microvesicle Analysis: Correlation between clinical outcomes and levels of circulating microvesicles.
  Serum Multiplex Panel: Correlation between clinical outcomes and serum biomarker levels (e.g., cytokines, chemokines), measured in concentration units (e.g., pg/mL).
Overall Survival (OS) | 2 years
  Time from treatment initiation to death from any cause, measured in months.
Progression-Free Survival (PFS) | 2 years
  Time from treatment initiation to disease progression or death, whichever occurs first, measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Camila MV Moniz, Doctor, Principal Investigator — Oncologist
Locations (8):
- Brazil (8):
  - DF Star, Brasília, Brasília
  - Hospital São Carlos, Fortaleza, Ceará
  - Hospital São Rafael, Salvador, Estado de Bahia
  - Hospital Santa Cruz, Curitiba, Paraná
  - IDOR Recife, Recife, Pernambuco
  - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro, Rio de Janeiro
  - Instituto D'or de Pesquisa e Ensino, São Paulo, São Paulo
  - Instituto do Câncer do Estado de São Paulo - ICESP, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No
It has been decided not to share individual participant data (IPD) related to the study for several reasons. Protecting the privacy of participants is a priority. Sharing IPD may expose sensitive information that, even when de-identified, can be traced back to individuals.
  Furthermore, the complexity of the data makes sharing challenging without the risk of misunderstandings or misinterpretations, which could compromise the integrity of the research. Sharing IPD without the explicit consent of participants may violate ethical principles of respect and protection.
  There is also a need to comply with regulatory guidelines governing data sharing to avoid potential legal issues. Finally, the focus will be on disseminating aggregated results that can benefit the scientific community and the public without compromising individual privacy.

REFERENCES:
- [Background] Bogaerts J, Sydes MR, Keat N, McConnell A, Benson A, Ho A, Roth A, Fortpied C, Eng C, Peckitt C, Coens C, Pettaway C, Arnold D, Hall E, Marshall E, Sclafani F, Hatcher H, Earl H, Ray-Coquard I, Paul J, Blay JY, Whelan J, Panageas K, Wheatley K, Harrington K, Licitra L, Billingham L, Hensley M, McCabe M, Patel PM, Carvajal R, Wilson R, Glynne-Jones R, McWilliams R, Leyvraz S, Rao S, Nicholson S, Filiaci V, Negrouk A, Lacombe D, Dupont E, Pauporte I, Welch JJ, Law K, Trimble T, Seymour M. Clinical trial designs for rare diseases: studies developed and discussed by the International Rare Cancers Initiative. Eur J Cancer. 2015 Feb;51(3):271-81. doi: 10.1016/j.ejca.2014.10.027. Epub 2014 Dec 24. PMID 25542058
- [Background] Cortes J, Kim SB, Chung WP, Im SA, Park YH, Hegg R, Kim MH, Tseng LM, Petry V, Chung CF, Iwata H, Hamilton E, Curigliano G, Xu B, Huang CS, Kim JH, Chiu JWY, Pedrini JL, Lee C, Liu Y, Cathcart J, Bako E, Verma S, Hurvitz SA; DESTINY-Breast03 Trial Investigators. Trastuzumab Deruxtecan versus Trastuzumab Emtansine for Breast Cancer. N Engl J Med. 2022 Mar 24;386(12):1143-1154. doi: 10.1056/NEJMoa2115022. PMID 35320644
- [Background] DuBois SG, Laetsch TW, Federman N, Turpin BK, Albert CM, Nagasubramanian R, Anderson ME, Davis JL, Qamoos HE, Reynolds ME, Cruickshank S, Cox MC, Hawkins DS, Mascarenhas L, Pappo AS. The use of neoadjuvant larotrectinib in the management of children with locally advanced TRK fusion sarcomas. Cancer. 2018 Nov 1;124(21):4241-4247. doi: 10.1002/cncr.31701. Epub 2018 Sep 11. PMID 30204247
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Li BT, Smit EF, Goto Y, Nakagawa K, Udagawa H, Mazieres J, Nagasaka M, Bazhenova L, Saltos AN, Felip E, Pacheco JM, Perol M, Paz-Ares L, Saxena K, Shiga R, Cheng Y, Acharyya S, Vitazka P, Shahidi J, Planchard D, Janne PA; DESTINY-Lung01 Trial Investigators. Trastuzumab Deruxtecan in HER2-Mutant Non-Small-Cell Lung Cancer. N Engl J Med. 2022 Jan 20;386(3):241-251. doi: 10.1056/NEJMoa2112431. Epub 2021 Sep 18. PMID 34534430
- [Background] Marabelle A, Fakih M, Lopez J, Shah M, Shapira-Frommer R, Nakagawa K, Chung HC, Kindler HL, Lopez-Martin JA, Miller WH Jr, Italiano A, Kao S, Piha-Paul SA, Delord JP, McWilliams RR, Fabrizio DA, Aurora-Garg D, Xu L, Jin F, Norwood K, Bang YJ. Association of tumour mutational burden with outcomes in patients with advanced solid tumours treated with pembrolizumab: prospective biomarker analysis of the multicohort, open-label, phase 2 KEYNOTE-158 study. Lancet Oncol. 2020 Oct;21(10):1353-1365. doi: 10.1016/S1470-2045(20)30445-9. Epub 2020 Sep 10. PMID 32919526
- [Background] Mok TSK, Wu YL, Kudaba I, Kowalski DM, Cho BC, Turna HZ, Castro G Jr, Srimuninnimit V, Laktionov KK, Bondarenko I, Kubota K, Lubiniecki GM, Zhang J, Kush D, Lopes G; KEYNOTE-042 Investigators. Pembrolizumab versus chemotherapy for previously untreated, PD-L1-expressing, locally advanced or metastatic non-small-cell lung cancer (KEYNOTE-042): a randomised, open-label, controlled, phase 3 trial. Lancet. 2019 May 4;393(10183):1819-1830. doi: 10.1016/S0140-6736(18)32409-7. Epub 2019 Apr 4. PMID 30955977
- [Background] Schmid P, Cortes J, Pusztai L, McArthur H, Kummel S, Bergh J, Denkert C, Park YH, Hui R, Harbeck N, Takahashi M, Foukakis T, Fasching PA, Cardoso F, Untch M, Jia L, Karantza V, Zhao J, Aktan G, Dent R, O'Shaughnessy J; KEYNOTE-522 Investigators. Pembrolizumab for Early Triple-Negative Breast Cancer. N Engl J Med. 2020 Feb 27;382(9):810-821. doi: 10.1056/NEJMoa1910549. PMID 32101663